CLINICAL TRIAL: NCT03751436
Title: Phase Ib/II Study of Enzalutamide With Venetoclax (ABT-199) in Patients With Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Brief Title: Enzalutamide With Venetoclax in Treating Patients With Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 63418; NCI-2018-02448 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 63418 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Metastatic Prostate Carcinoma in the Soft Tissue; Prostate Carcinoma Metastatic in the Bone; PSA Progression; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (venetoclax, enzalutamide) (Experimental): Patients receive venetoclax PO QD and enzalutamide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide; Drug: Venetoclax

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of venetoclax when given together with enzalutamide and to see how well they work in treating patients with castration resistant prostate cancer that has spread to other places in the body. Androgens can cause the growth of prostate cancer cells. Drugs, such as enzalutamide, may lessen the amount of androgens made by the body. Venetoclax may target a special group of prostate cancer cells that is known to lead to resistance to treatment. Giving enzalutamide and venetoclax may work better in treating patients with castration resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD), and recommended phase II dose (RP2D) of enzalutamide in combination with venetoclax in patients with metastatic castrate resistant prostate cancer (mCRPC). (Phase Ib)
* To characterize the safety and tolerability profile of enzalutamide in combination with venetoclax in patients with metastatic castrate resistant prostate cancer (mCRPC). (Phase Ib)
* To evaluate the efficacy of venetoclax in combination with enzalutamide in patients with metastatic castrate resistant prostate cancer (mCRPC) that are enzalutamide-naive, as measured by 12-month progression free survival rate. (Phase II)

SECONDARY OBJECTIVES:

* To assess PSA50 response as well as circulating tumor cell (CTC) response in patients who received venetoclax + enzalutamide. (Phase II)

  -To estimate the proportion of patients who received venetoclax + enzalutamide and remain radiographic progression free at 6 months. (Phase II)
* To estimate the time to first skeletal-related event (SRE) and the time to first symptomatic skeletal event (SSE). (Phase II)

  - To estimate the time to clinical progression. (Phase II)
* To estimate the time to initiation of new systemic treatment for prostate cancer. (Phase II)
* Assess the effect of venetoclax + enzalutamide on overall survival. (Phase II)

PHARMACOKINETIC OBJECTIVES:

I. To characterize the pharmacokinetic (PK) profiles of enzalutamide and venetoclax when given in combination to patients with metastatic castrate resistant prostate cancer (mCRPC).

II. Comprehensive analyses of venetoclax levels to assure that they are in the therapeutic range.

EXPLORATORY BIOMARKER OBJECTIVES:

I. To identify non-inherited biomarkers that are predictive of response to study treatment (i.e., predictive biomarkers), are associated with progression to a more severe disease state (i.e., prognostic biomarkers), are associated with acquired resistance to study treatment, are associated with susceptibility to developing adverse events, can provide evidence of study treatment activity, can increase the knowledge and understanding of prostate cancer biology or study treatment mechanism of action, or can contribute to improvement of diagnostic assays.

OUTLINE: This is a phase Ib, dose-escalation study of venetoclax followed by a phase II study.

Patients receive venetoclax orally (PO) once daily (QD) and enzalutamide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of diagnosis of prostate cancer.
* Documented progressive metastatic castrate resistant prostate cancer (mCRPC) based on at least one of the following criteria:

  * Prostate specific antigen (PSA) progression defined as 25% increase over baseline value with an increase in the absolute value of at least 2 ng/mL that is confirmed by another PSA level with a minimum of a 1 week interval and a minimum PSA of 2 ng/mL.
  * Soft-tissue progression defined as an increase >= 20% in the sum of the longest diameter (LD) of all target lesions based on the smallest sum LD since treatment started or the appearance of one or more new lesions.
  * Progression of bone disease (evaluable disease) or, new bone lesion(s), by bone scan.
  * If on an anti-androgen, must have documented progression 6 weeks after stopping anti-androgen therapy.
* Willing to undergo a biopsy, if readily available biopsy site present (i.e., nodal or visceral metastasis).
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
* Have testosterone level of < 50 ng/dL. Note: Patients must continue primary androgen deprivation with a luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist) if they have not undergone orchiectomy.
* White blood cells >= 1.5 x 10^9/L (obtained within 14 days prior to treatment start)
* Platelets (UNVPLT) >= 100 x 10^9/L (obtained within 14 days prior to treatment start)
* Hemoglobin (HGB) >= 9 g/dL (obtained within 14 days prior to treatment start)
* Potassium (K), total calcium (CA) (corrected for serum albumin), magnesium, sodium (NA) and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication (obtained within 14 days prior to treatment start)
* Total calcium (CA) (corrected for serum albumin) within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication (obtained within 14 days prior to treatment start)
* Magnesium within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication (obtained within 14 days prior to treatment start)
* Sodium (NA) within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication (obtained within 14 days prior to treatment start)
* Phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication (obtained within 14 days prior to treatment start)
* Institutional normalized ratio (INR) =< 1.5 (obtained within 14 days prior to treatment start)
* Adequate renal function as demonstrated by a creatinine clearance >= 30 mL/min; calculated by the Cockcroft Gault formula
* Aspartate aminotransferase (aspartate transaminase [AST]) and alanine aminotransferase (alanine transaminase [ALT]) =< 3 X upper limit of normal (ULN). If the patient has liver metastases, ALT and AST must still be =< 3 x ULN. Patients with liver metastases and AST/ALT above this limit will not be enrolled (obtained within 14 days prior to treatment start)
* Total serum bilirubin =< 1.5 x ULN (unless bilirubin rise is due to Gilbert?s syndrome or of non-hepatic origin); or total bilirubin (TBILI) =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert?s syndrome (obtained within 14 days prior to treatment start)
* Ability to swallow and retain oral medication (without crushing, dissolving or chewing tablets).
* Phase Ib only: Prior enzalutamide treatment and/or other approved treatments for CRPC are acceptable
* Phase II only: Participants MUST be treatment naive in the CRPC setting: i.e., no prior exposure to abiraterone acetate other specific CYP-17 inhibitors; no prior exposure to enzalutamide or investigational androgen receptor (AR) targeted agents; and no prior exposure to chemotherapy and or RAD-223.
* Sexually active males must agree to use a condom during intercourse while taking the study drug and for at least 3 months after stopping study treatment. Sexually active males should not father a child during this period. A condom is required to be used by vasectomized men in order to prevent delivery of the drug via seminal fluid. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.
* Participant or legal representative must understand the investigational nature of this study and voluntarily sign and date an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Phase II only: Prior exposure to abiraterone acetate.
* Phase II only: Prior exposure to BCL-2 inhibitors agents like venetoclax.
* Phase II only: Prior chemotherapy for castration resistant disease. Chemotherapy given in the castration-sensitive setting is permissible if stopped at least 4 weeks prior to treatment start.
* Phase II only: Prior isotope therapy with strontium-89, samarium or radium-223 within 12 weeks of treatment start.
* Subject has acute promyeloctyic leukemia
* Subject has known active CNS involvement with AML
* Participants with known symptomatic brain metastases.
* Participant has a concurrent malignancy or malignancy within 3 years of treatment start, with the exception of adequately treated, basal or squamous cell carcinoma, nonmelanomatous skin cancer or curatively resected cervical cancer.
* Participant has a known history of human immunodeficiency virus (HIV) infection (testing not mandatory);
* Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate
* Uncontrolled and/or active systemic infection (viral, bacterial or fungal).
* Participant has clinically significant, uncontrolled heart disease and/or recent events including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, uncontrolled hypertension, uncontrolled arrhythmia, stroke, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to treatment start
  * Cardiac history of CHF requiring treatment or Ejection fraction ≤ 50% or chronic stable angina
  * A cardiovascular disability status of New York Heart Association Class > 2
  * Class 2 is - Defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea or angina pain
  * On screening 12 lead electrocardiography (ECG), any of the following cardiac parameters: bradycardia (heart rate < 50 at rest), tachycardia (heart rate > 90 at rest), PR interval > 220 msec, QRS interval > 109 msec or, Fridericia's correction formula (QTcF) > 450 msec. Congenital long QT syndrome or family history of long QT syndrome.
* DLCO <=65% or FEVI <= 65&
* Treatment with any of the following within 7 days prior to the first dose of study drug:

  * Steroid therapy for anti-neoplastic intent
  * Moderate or strong cytochrome P450 3A (CYP3A) inhibitors
  * Moderate or strong CYP3A inducers
  * Medications that have a known risk to prolong the QT interval or induce Torsades de Pointes
  * Herbal preparations/medications
* Participants receiving any medications or substances that are inhibitors or inducers of CYP2C8 enzymes are ineligible.
* Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

  * Grapefruit or grapefruit products
  * Seville oranges (including marmalade containing Seville oranges)
  * Star fruit.
* Patient who has received radiotherapy =< 4 weeks prior to start of treatment or limited field radiation for palliation =< 2 weeks prior to treatment start and, who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom >= 30% of the bone marrow was irradiated.
* Patients with central nervous system (CNS) involvement.
* Patients with seizure disorder.
* Patient has not recovered from all toxicities related to prior anticancer therapies to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0) grade < =1 (Exception to this criterion: patients with any grade of alopecia are allowed to enter the study).
* Participant has any other concurrent severe and/or uncontrolled medical condition that would cause, in the investigator's judgment, an unacceptable safety risk.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase Ib) | Up to 28 days
  The MTD will be determined based on the rate of dose-limiting toxicities (DLTs). Adverse events will be categorized and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Recommended phase 2 dose (RP2D) (Phase Ib) | Up to 28 days
  Will be selected based on the overall tolerability of the regimen, but will not exceed the MTD.
Progression free survival (Phase II) | Time from start of treatment combination therapy to disease progression, assessed at 12 months
  Prostate Cancer Working Group (PCWG)3 will be used to evaluate PSA response and progression as well as progression on bone scans. Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 will be used to assess response and progression for nodal and visceral metastasis. The Kaplan-Meier product-limit estimator will be used.

SECONDARY OUTCOMES:
PSA50 (Phase II) | Up to 3 years
  Will be defined as the proportion of patients with a >= 50% reduction in PSA from baseline.
Circulating tumor cell (CTC) conversion in patients who enter the trial with unfavorable CTCs (five or more cells per 7.5 mL of blood) (Phase II) | Up to 3 years
  Conversion to favorable status is defined as four or fewer cells per 7. mL of blood.
Radiographic (r)PFS (Phase II) | Time from day (D) 1 of treatment to the date when the first site of disease is found to progress (using a manifestation-specific definition off progression), or death, whichever occurs first, assessed up to 3 years
  Will be defined per PCWG3.
Proportion of patients who remain radiographic progression free defined per PCWG3 (Phase II) | Tt 6 months
Overall response rate (ORR) (Phase II) | Up to 3 years
  For patients with measurable soft tissue disease, ORR will be defined as the proportion of patients with a complete response (CR) or partial response (PR) per PCWG3.
Duration of response (DOR) (Phase II) | From the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that radiographic progression is documented per PCWG3, assessed up to 3 years
Time to first skeletal-related event (SRE) (Phase II) | Time from D1 of treatment to the date of first SRE, assessed up to 3 years
Time to clinical progression (Phase II) | Time from D1 of treatment to the date of clinical progression, assessed up to 3 years
Time to initiation of new systemic treatment for prostate cancer (Phase II) | Time from D1 of treatment to the date any new systemic treatment for prostate cancer is initiated, assessed up to 3 years
Overall survival (Phase II) | From the time of initiation of the combination therapy until death from any cause, assessed up to 3 years
  The Kaplan-Meier product-limit estimator will be used.

OTHER OUTCOMES:
Observed serum concentration of enzalutamide | Up to 3 years
  Pharmacokinetic (PK) parameters will include: area under the concentration versus time curves (AUC)
Observed serum concentration of venetoclax | Up to 3 years
  PK parameters will include: area under the concentration versus time curves (AUC)
Biomarker analysis | Up to 3 years
  Tumor and blood samples will be assessed. Will be summarized using standard descriptive statistics.
Observed serum concentration of venetoclax | Up to 3 years
  PK parameters will include: Maximum concentration (Cmax)
Observed serum concentration of venetoclax | Up to 3 years
  PK parameters will include: time to maximum concentration (Tmax)
Observed serum concentration of venetoclax | Up to 3 years
  PK parameters will include minimum (trough) concentration (Ctrough)
Observed serum concentration of venetoclax | Up to 3 years
  PK parameters will include elimination half-life (T1/2)
Observed serum concentration of venetoclax | Up to 3 years
  PK parameters will include volume of distribution (Vd)/bioavailability or fraction absorbed (F), clearance (CL)/F
Observed serum concentration of venetoclax | Up to 3 years
  PK parameters will include peak-to-trough ratio
Observed serum concentration of venetoclax | Up to 3 years
  PK parameters will include accumulation ratio
Observed serum concentration of enzalutamide | Up to 3 years
  PK parameters will include maximum concentration (Cmax)
Observed serum concentration of enzalutamide | Up to 3 years
  PK parameters will include time to maximum concentration (Tmax)
Observed serum concentration of enzalutamide | Up to 3 years
  PK parameters will include minimum (trough) concentration (Ctrough)
Observed serum concentration of enzalutamide | Up to 3 years
  PK parameters will include elimination half-life (T1/2)
Observed serum concentration of enzalutamide | up to 3 years
  PK parameters will include volume of distribution (Vd)/bioavailability or fraction absorbed (F), clearance (CL)/F
Observed serum concentration of enzalutamide | Up to 3 years
  PK parameters will include peak-to-trough ratio
Observed serum concentration of enzalutamide | Up to 3 years
  PK parameters will include accumulation ratio

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal Chatta, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Perimbeti S, Jamroze A, Gopalakrishnan D, Jain R, Jiang C, Holleran JL, Parise RA, Bies R, Quinn D, Attwood K, Liu X, Green K, Kirk JS, Beumer JH, Tang DG, Chatta G. Phase Ib study of enzalutamide with venetoclax in patients with metastatic castration-resistant prostate cancer. Cancer Chemother Pharmacol. 2025 Nov 29;95(1):115. doi: 10.1007/s00280-025-04840-2. PMID 41315064
- [Derived] Rodriguez Y, Unno K, Truica MI, Chalmers ZR, Yoo YA, Vatapalli R, Sagar V, Yu J, Lysy B, Hussain M, Han H, Abdulkadir SA. A Genome-Wide CRISPR Activation Screen Identifies PRRX2 as a Regulator of Enzalutamide Resistance in Prostate Cancer. Cancer Res. 2022 Jun 6;82(11):2110-2123. doi: 10.1158/0008-5472.CAN-21-3565. PMID 35405009